CLINICAL TRIAL: NCT04966403
Title: Distinct Effects of Trampoline-based Stretch-shortening Cycle Exercises on Muscle Strength and Postural Control in Children With Down Syndrome: A Randomized Controlled Study
Brief Title: Effects of Stretch-shortening Cycle Exercises Postural Control in Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Collaborators: Cairo University (Other); Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Maged Basha, Principal Investigator, Assistant Professor, College of Medical Rehabilitation, Qassim University, Saudi Arabia. Consultant Physical Therapist, El-Sahel Teaching Hospital, General Organization for Teaching Hospitals and Institutes, Cairo, Egypt., Qassim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0018/0086
Record Dates: First submitted 2021-07-14; First posted 2021-07-19 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome | interventions — Physical Fitness; Postural Balance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard physical therapy (Experimental): Participants in the standard physical therapy received the standard physical therapy (sPT) program, which was conducted according to the needs of each participant and was generally concerned with building strength, enhancing developmental skills, boosting balance, coordination, and postural control, improving physical fitness, and minimizing the development of the compensatory movement patterns that children with DS are likely to develop.
  Interventions: Other: Standard physical therapy
- trampoline-based stretch-shortening cycle exercises (Experimental): In addition to the sPT, the SSC group received 15-minute SSC exercise sessions, twice weekly, with a total of 24 sessions over 12 successive weeks.
  Interventions: Other: trampoline-based stretch-shortening cycle exercises

INTERVENTIONS:
Other: Standard physical therapy — building strength, enhancing developmental skills, boosting balance, coordination, and postural control
  Other Names: physical fitness
  Arms: standard physical therapy
Other: trampoline-based stretch-shortening cycle exercises — muscle strength
  Other Names: postural control
  Arms: trampoline-based stretch-shortening cycle exercises

SUMMARY:
To investigate the effect of a 3-month, trampoline-based stretch-shortening cycle (SSC) exercises on muscle strength and postural control in children with Down syndrome.

DETAILED DESCRIPTION:
a variety of physical therapy techniques are being used to improve lower limb muscle strength and postural control in children with Down syndrome including, but not limited to, progressive resistance training, hippotherapy, aquatic therapy, and isokinetic strength training. Stretch-shortening (SSC) exercises-also referred to as plyometric exercises, is a traditional form of resistance training that involves three-phase muscle contraction during dynamic movements (like jumping and hopping), where the muscle moves rapidly through the eccentric, isometric, and concentric phases.

ELIGIBILITY:
Inclusion Criteria:

* age between 7 and 9 years.
* able to follow one step motor commands.
* independent ambulators.
* not suffering from atlantoaxial joint instability as reported from their medical files.

Exclusion Criteria:

* Children with un-corrected cardiac anomalies.
* Children with un-corrected vision or hearing loss.
* Children with un-corrected pulmonary disorders.
* Children with un-corrected neurological signs as epilepsy.
* Children who had a history of musculoskeletal surgery in the lower extremities through the past year.

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
Grade of Muscle strength by hand-held dynamometer | at baseline
  A calibrated hand-held dynamometer (Micro FET2, Hoggan Health Technologies Inc., UT, USA) was used
Grade of Muscle strength by hand-held dynamometer | after 12 weeks
  A calibrated hand-held dynamometer (Micro FET2, Hoggan Health Technologies Inc., UT, USA) was used

SECONDARY OUTCOMES:
Postural control index by Balance Biodex System | at baseline
  Postural stability indices were assessed through the Balance Biodex System (Biodex Medical Systems, Shirley, NY),
Postural control index by Balance Biodex System | after 12 weeks
  Postural stability indices were assessed through the Balance Biodex System (Biodex Medical Systems, Shirley, NY),

CONTACTS AND LOCATIONS:
Overall Officials: Alshimaa Azab, PhD, Study Director — Cairo University
Locations (1):
- King Khalid Hospital, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study is available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.

REFERENCES:
- [Background] Alsakhawi RS, Elshafey MA. Effect of Core Stability Exercises and Treadmill Training on Balance in Children with Down Syndrome: Randomized Controlled Trial. Adv Ther. 2019 Sep;36(9):2364-2373. doi: 10.1007/s12325-019-01024-2. Epub 2019 Jul 12. PMID 31301057
- [Result] Aalizadeh B, Mohammadzadeh H, Khazani A, Dadras A. Effect of a Trampoline Exercise on the Anthropometric Measures and Motor Performance of Adolescent Students. Int J Prev Med. 2016 Jul 13;7:91. doi: 10.4103/2008-7802.186225. eCollection 2016. PMID 27512557
- [Result] Champagne D, Dugas C. Improving gross motor function and postural control with hippotherapy in children with Down syndrome: case reports. Physiother Theory Pract. 2010 Nov;26(8):564-71. doi: 10.3109/09593981003623659. Epub 2010 Jul 31. PMID 20673078